CLINICAL TRIAL: NCT00215423
Title: Study in Patients With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Director, Clinical Affairs, Dey
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DL-057
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2008-08

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Formoterol Fumarate; Formoterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

INTERVENTIONS:
Drug: Formoterol Fumarate

SUMMARY:
The purpose of this study is to determine which dose of the investigational drug is the most safe and effective for the treatment of COPD compared to the control drug

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* History of cigarette smoking

Exclusion Criteria:

* Clinical diagnosis of asthma
* Significant pulmonary disease other than COPD
* Other significant major organ disease(s)

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49
Dates: Primary Completion 2003-12 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Measure of lung function

SECONDARY OUTCOMES:
Change in lung function, as well as vital signs
Physical Exam results, adverse event reporting, etc

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Research Site, Phoenix, Arizona
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Hines, Illinois
  - Research Site, Shawnee Mission, Kansas
  - Research Site, Butte, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Medford, Oregon

REFERENCES:
- [Result] Gross NJ, Kerwin E, Levine B, Kim KT, Denis-Mize K, Hamzavi M, Carpenter M, Rinehart M. Nebulized formoterol fumarate: Dose selection and pharmacokinetics. Pulm Pharmacol Ther. 2008 Oct;21(5):818-23. doi: 10.1016/j.pupt.2008.07.002. Epub 2008 Jul 8. PMID 18655841